CLINICAL TRIAL: NCT00000987
Title: A Phase I Study of Combination Chemotherapy (Adriamycin, Bleomycin, and Vincristine) and Azidothymidine in the Treatment of AIDS Related Kaposi's Sarcoma
Brief Title: A Study of Chemotherapy Plus Azidothymidine in the Treatment of Kaposi's Sarcoma in Patients With AIDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 075; 11049 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Vincristine; Doxorubicin; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Bleomycin
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Bleomycin; Vincristine; Doxorubicin; Zidovudine

INTERVENTIONS:
Drug: Bleomycin sulfate
Drug: Vincristine sulfate
Drug: Doxorubicin hydrochloride
Drug: Zidovudine

SUMMARY:
To study the safety and maximum tolerated dose (MTD) of combined chemotherapy when it is administered to patients with advanced Kaposi's sarcoma together with one of two different doses of zidovudine (AZT).

The combination of AZT and chemotherapy may be effective in treating the tumor as well as preventing the life-threatening infections when used for patients with AIDS and Kaposi's sarcoma. The MTD of combined chemotherapy is being determined so that the information will be available for future studies, when the relative effectiveness of the two doses of AZT has been learned.

DETAILED DESCRIPTION:
The combination of AZT and chemotherapy may be effective in treating the tumor as well as preventing the life-threatening infections when used for patients with AIDS and Kaposi's sarcoma. The MTD of combined chemotherapy is being determined so that the information will be available for future studies, when the relative effectiveness of the two doses of AZT has been learned.

AMENDED: AZT by mouth. If the treatment is well tolerated, subsequent groups of patients are started on increasing doses of doxorubicin combined with the same dose of bleomycin and vincristine. After determination of the MTD of chemotherapy in combination with AZT, the 2nd phase begins in which AZT is given and the first group of patients is given bleomycin and vincristine only. If this combination is well tolerated, then the subsequent groups are started on increasing doses of doxorubicin with the same dose of bleomycin, vincristine and AZT. The MTD of chemotherapy in combination with AZT is then determined. Patients achieving maximum response to the tumor are maintained on AZT alone. This is an outpatient study, and patients are seen every 2 weeks for evaluation, with a physical examination every month. Original design: The combination of chemotherapy and AZT is given to groups of four patients each, the first group beginning with bleomycin and vincristine, without the addition of doxorubicin. The chemotherapy is given intravenously every 2 weeks. This is combined first with AZT by mouth.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Medication for grades 1 and 2 oral toxicity. Antiemetic agents, except steroids, for gastrointestinal toxicity. Toxicity grades according to NIAID Recommendations for Grading of Acute and Subacute Toxic Effects (Adults).

Patients must demonstrate any of the following clinical and laboratory findings:

* 25 or more mucocutaneous lesions with or without lymphedema.
* Progressive Kaposi's sarcoma (KS) with 10 or more new lesions in the month prior to study entry or visceral involvement.
* Oral mucosal lesion(s) requiring therapy.
* Prior history of Pneumocystis carinii pneumonia (PCP) or Mycobacterium avium intracellulare.

Patients with any of the following constitutional symptoms with no etiology established may be included:

* Temperature > 38 degrees C and/or drenching night sweats for more than 1 month.
* Watery diarrhea (= or > 3 stools/day) for 2 or more weeks.
* Weight loss > 10 percent of normal. Patients with carcinoma in situ of the cervix or localized squamous or basal cell carcinoma of the skin may be included.

Active alcohol or drug abuse sufficient to prevent adequate compliance with study therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions will be excluded:

* Peripheral sensory or motor neuropathy.
* Opportunistic infections requiring therapy.
* Significant pulmonary (exertional dyspnea with minimal exercise) or cardiac insufficiency (New York Heart Association, status > 2).
* Serious neuropsychiatric illness which would prevent informed consent of intensive treatment.

Concurrent Medication:

Excluded:

* Any drugs causing anemia, neutropenia, or significant risk of nephrotoxicity. Patients with a history of other systemic malignancies or lymphomas, except carcinoma in situ of the cervix or localized squamous or basal cell carcinoma of the skin, will be excluded from the study.

Prior Medication:

Excluded:

* Systemic antineoplastic chemotherapy.
* Excluded within 30 days of study entry:
* Any other investigational therapy.
* Antiretroviral agents (zidovudine, ribavirin).
* Immunomodulating agents (steroids, interferons, naltrexone, isoprinosine, and interleukin-2).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Study Completion 1992-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: PS Gill, Study Chair; S Miles, Study Chair
Locations (1):
- UCLA CARE Center CRS, Los Angeles, California, United States

REFERENCES:
- [Background] Brambilla D, Coombs R, Bremer JW, Reichelderfer PS, Kalish L, Shapiro DE. The contributions of assay variation and biological variation to the variability of HIV RNA measurements in serially collected clinical specimens. Int Conf AIDS. 1998;12:805 (abstract no 42163)
- [Background] Gill PS, Miles SA, Mitsuyasu RT, Montgomery T, McCarthy S, Espina BM, Feldstein M, Levine AM. Phase I AIDS Clinical Trials Group (075) study of adriamycin, bleomycin and vincristine chemotherapy with zidovudine in the treatment of AIDS-related Kaposi's sarcoma. AIDS. 1994 Dec;8(12):1695-9. doi: 10.1097/00002030-199412000-00009. PMID 7534090